CLINICAL TRIAL: NCT00924183
Title: Measuring Response to Depression Treatment: A Study Comparing the Sensitivity of Multiple Outcome Measures to Change
Brief Title: Measuring Response to Depression Treatment
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Dr. D McIntosh & Dr. K Kjernisted Clinical Research Inc. (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Dr. Diane McIntosh, Dr. D McIntosh & Dr. K Kjernisted Clinical Research Inc.
Other Study IDs: D1443L00014
Record Dates: First submitted 2009-06-10; First posted 2009-06-18 (Estimated); Last update posted 2011-03-23 (Estimated); Status verified 2011-03

CONDITIONS: Depression
Keywords: Depression; Symptom scales; Symptom measures; Vancouver Semi-Structured Interview for Depression; V-SID; VSID; treatment-as-usual; treatment as usual; open-label; open label; Major Depressive Episode; MDE
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and white blood cells will be isolated from whole blood samples and will be stored for future analysis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Treatment-as-usual: All patients will receive treatment as usual: antidepressant medication and/or cognitive behavioral therapy (CBT). Patients' results will be compare to their own baseline measurements.
  Interventions: Other: Treatment-as-usual

INTERVENTIONS:
Other: Treatment-as-usual

SUMMARY:
The primary goal of this study is to compare a new symptoms rating questionnaire, called the Vancouver Semi-Structured Interview for Depression (V-SID), to the traditionally used questionnaires. The investigators predict that the V-SID will be more sensitive to patients' improvement than are traditional questionnaires.

DETAILED DESCRIPTION:
Depression is sometimes associated with difficulties in thinking skills. Recent evidence suggests that in those people who have thinking difficulties, effective treatment and improvement of depression can also result in improved thinking skills. Therefore, a test of thinking skills is included in this study.

This study will also evaluate three other potential indicators of treatment response: cortisol, cytokines, and grip strength.

ELIGIBILITY:
Inclusion Criteria:

* Major depressive episode, diagnosed using the Mini-International Neuropsychiatric Interview (MINI)
* Depression not currently effectively treated
* Age 19 to 65 years

Exclusion Criteria:

* Co-morbid Axis I disorders (co-morbid anxiety symptoms, including generalized anxiety or panic attacks, are not exclusionary if they are present in the context of a primary mood disorder)

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects will diagnosed with a current major depressive episode. They will be recruited from a community healthcare centre.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2008-06; Primary Completion 2011-07 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Hamilton Rating Scale for Depression (HAM-D) | Pre-Baseline, Day 0, Week 1, Week 4, Week 8
Vancouver Semi-Structured Interview for Depression (V-SID) | Pre-Baseline, Day 0, Week 1, Week 4, Week 8
Montgomery-Asberg Depression Rating Scale (MADRS) | Pre-Baseline, Day 0, Week 1, Week 4, Week 8
Clinical Global Impression | Pre-Baseline, Day 0, Week 1, Week 4, Week 8, Followup
Hamilton Rating Scale for Anxiety (HAM-A) | Pre-Baseline, Day 0, Week 1, Week 4, Week 8
British Columbia Major Depression Inventory (BC-MDI) | Pre-Baseline, Day 0, Week 1, Week 4, Week 8
Quality of Life Enjoyment Satisfaction Questionnaire (Q-LES-Q) | Day 0, Week 8

SECONDARY OUTCOMES:
CNS Vital Signs | Pre-Baseline, Day 0, Week 8
British Columbia Cognitive Complaints Inventory (BC-CCI) | Pre-Baseline, Day 0, Week 1, Week 4, Week 8
Grip strength | Pre-Baseline, Day 0, Week 8
Cortisol level | Day 0, Week 8
Neuroimmunobiologic markers | Pre-Baseline, Week 8
Evaluation for Metabolic Syndrome | Day 0, Week 8, Followup

CONTACTS AND LOCATIONS:
Overall Officials: Diane McIntosh, MD, FRCPC, Principal Investigator — Dr. D McIntosh & Dr. K Kjernisted Clinical Research Inc.
Locations (1):
- Copeman Neuroscience Centre, Vancouver, British Columbia, Canada